CLINICAL TRIAL: NCT03301688
Title: A Similar Phase I Study on the Pharmacokinetics and Safety of Single-dose and Parallel Comparisons in Patients With Advanced NSCLC Treated With Recombinant Humanized Anti-PD-1 Monoclonal Antibody (JS001) Before and After Process Change
Brief Title: The Pharmacokinetics and Safety of Single-dose and Parallel Comparisons in Patients With NSCLC Treated With JS001
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Junshi Bioscience Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Junshi-JS001-012
Record Dates: First submitted 2017-09-29; First posted 2017-10-04 (Actual); Last update posted 2020-09-30 (Actual); Status verified 2020-09

CONDITIONS: NSCLC
Keywords: PD-1 antibody; phase 1 trial
MeSH Terms: interventions — toripalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A group (JS001 20161002) (Experimental): The subjects of A group will use 3 mg/kg doses every 2 weeks.Drug batch number is 20161002.
  Interventions: Biological: Toripalimab
- B group (JS001 20161108) (Experimental): The subjects of B group will use 3 mg/kg doses every 2 weeks.Drug batch number is 20161108.
  Interventions: Biological: Toripalimab

INTERVENTIONS:
Biological: Toripalimab — To compare the different drug batch number with different process
  Other Names: JS001, TAB001

SUMMARY:
This study was designed to evaluate the similarity of single-dose and parallel comparisons of recombinant humanized anti-PD-1 monoclonal antibody injections before and after process changes. It is designed to be a single-center, open and parallel controlled phase I study. Patients with advanced NSCLC will be enrolled.

After determining that the patient is qualified, the patient will be assigned to a batch of drug use in the order in which they are selected. The dosage of drug was set at 3 mg / kg. Planned to recruit subjects each 12 patients (24 cases) to participate in this study, taking into account a 20% dropout rate, so that the total of 15 patients (30 patients) subjects in each group in this study.

This study was divided into study phase (single-dose period) and follow-up stage (multiple-dose period).Each subject first conducted a single dose safety and pharmacokinetics (PK) study.If the subject did not develop adverse events that had significant clinical significance as suggested by the investigators within 28 days of the single dose and continued reorganization of the humanized anti-PD-1 monoclonal antibody injection to benefit the patient , and with the agreement of subjects, the subject will enter the follow-up phase (multiple-dose period). The same dose of recombinant humanized anti-PD-1 monoclonal antibody injection was administered once every 2 weeks and 4 consecutive cycles of treatment for one cycle of continuous period.Until the patient has developed tumor progression or an untolerated toxic side effect, the patient voluntarily exits the study or believes that the situation is not suitable for continuing treatment. There are follow-up of 90 days after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female aged 18 to 70 years are eligible;
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1
* Histologic diagnosis of NSCLS. Have failed at least 1 prior routine regimen for metastatic disease, or failed to tolerate the toxicity, or lack of any routine regimens.
* Providing with tumor specimen (for testing the expression of PD -L1 and the infiltrating lymphocytes);
* At least 1 measurable lesion (only 1 measurable lymph node lesion is excluded) (routine CT scan >=20mm, spiral CT scan >=10mm, no prior radiation to measurable lesions) Predicted survival >=6 months;
* Brain or meningeal metastases must be disposed with surgery or radiation, and be stable clinically for at least 8 weeks (prior systemic steroids was allowed, but concurrent administration of systemic steroids with the study drug is excluded).
* Screening laboratory values must meet the following criteria（within past 14 days）:

hemoglobin ≥ 9.0 g/dL neutrophils ≥ 1500 cells/ µL platelets ≥ 100 x 10^3/ µL total bilirubin ≤ 1.5 x upper limit of normal (ULN) aspartic transaminase (AST) and alanine transaminase (ALT) ≤ 2.5 x ULN without, and ≤ 5 x ULN with hepatic metastasis serum creatinine ≤1╳ULN，creatinine clearance >50ml/min (Cockcroft-Gault equation)

* Without systemic steroids within past 4 weeks
* Males or female of childbearing potential must: agree to use using a reliable form of contraception (eg, oral contraceptives, intrauterine device, control sex desire, double barrier method of condom and spermicidal) during the treatment period and for at least 12 months after the last dose of study drug.
* Must have read, understood, and provided written informed consent voluntarily. - Willing to adhere to the study visit schedule and the prohibitions and restrictions specified in this protocol.

Exclusion Criteria:

* Hypersensitivity to recombinant humanized anti-PD-1 monoclonal Ab or its components.
* Prior treatment with mAb within past 3 months (locally administration excluded)
* Prior antitumor therapy (including corticosteroids and immunotherapy) or participation in other clinical trials within past 4 weeks, or have not recovered from toxicities since the last treatment;
* Pregnant or nursing
* Abnormal Blood coagulation
* Positive tests for HIV, HCV, HBsAg or HBcAb with positive test for HBV DNA (>500IU/ml)
* History with pulmonary tuberculosis;
* Patients with any active autoimmune disease or a documented history of autoimmune disease, or history of syndrome that required systemic steroids or immunosuppressive medications, such as hypophysitis, pneumonia, colitis, hepatitis, nephritis, hyperthyroidism or hypothyroidism.
* Severe, uncontrolled medical condition that would affect patients' compliance or obscure the interpretation of toxicity determination or adverse events, including active severe infection, uncontrolled diabetes, angiocardiopathy (heart failure > class II NYHA, heart block >II grade, myocardial infarction, unstable arrhythmia or unstable angina within past 6 months, cerebral infarction within past 3 months) or pulmonary disease ( interstitial pneumonia, obstructive pulmonary disease or symptomatic bronchospasm).
* Prior treatment with bone marrow stimulating factors，such as CSF (colony stimulating factor), EPO (erythropoietin), within past 1 weeks
* Prior live vaccine therapy within past 4 weeks.
* Prior major surgery within past 4 weeks (diagnostic surgery excluded).
* Psychiatric medicines abuse without withdrawal, or history of psychiatric illness.
* Prior malignancy active within the previous 5 years except for locally curable cancers that have been apparently cured, such as basal cell skin cancer or carcinoma in situ of the cervix.
* Underlying medical condition that, in the Investigator's opinion, would increase the risks of study drug administration or obscure the interpretation of toxicity determination or adverse events.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2017-09-18 (Actual); Primary Completion 2018-09-15 (Actual); Study Completion 2019-12-15 (Actual)

PRIMARY OUTCOMES:
Area Under the Curve (AUC) after single dose injection of Anti-PD-1 mAb | 6 months

SECONDARY OUTCOMES:
Objective response rate (ORR) | 6 months
  Objective Response Rate (ORR) by irRC and RECIST 1.1
Duration of response (DOR) | 6 months
  Duration of response (DOR) by irRC and RECIST 1.1
Disease control rate (DCR) | 6 months
  Disease control rate (DCR) by irRC and RECIST 1.1
Progression Free Survival (PFS) | 6 months
  Progression Free Survival (PFS) by irRC and RECIST 1.1
Overall Survival (OS) | 6 months
  Overall Survival (OS) by irRC and RECIST 1.1
Time to response (TTR) | 6 months
  Time to response (TTR) by irRC and RECIST 1.1
Maximum Plasma Concentration (Cmax) after single dose injection of Anti-PD-1 Monoclonal Antibody (mAb) | 6 months
Peak Time (Tmax) after single dose injection of Anti-PD-1 mAb | 6 months
t1/2 after single dose injection of Recombinant Humanized Anti-PD-1 mAb | 6 months
Plasma clearance (CL) after single dose injection of Anti-PD-1 mAb | 6 months
Apparent volume of distribution (V) after single dose injection of Anti-PD-1 mAb | 6 months
Minimum Plasma Concentration (Cmin) of steady state after multiple dose injection of Anti-PD-1 mAb | 6 months
Average Plasma Concentration (Cav) of steady state after multiple dose injection of Anti-PD-1 mAb | 6 months
degree of fluctuation (DF) of steady state after multiple dose injection of Anti-PD-1 mAb | 6 months
Apparent volume of distribution of steady state (Vss) after multiple dose injection of Anti-PD-1 mAb | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jie Wang, MD, PhD, Principal Investigator — Cancer Hospital Chinese Academy of Medical Science
Locations (1):
- Cancer Hospital Chinese Academy of Medical Science, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided